CLINICAL TRIAL: NCT00630227
Title: Phase 2 Study of the 20 mL Biologic Lung Volume Reduction (BLVR) System in Patients With Homogeneous or Upper Lobe Predominant Emphysema
Brief Title: Biologic Lung Volume Reduction (BLVR) Phase 2 Homogeneous Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-C07-002
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Homogeneous Emphysema
Keywords: emphysema; chronic obstructive pulmonary disease; lung volume reduction
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): all patients are treated with the experimental therapy
  Interventions: Biological: Biologic Lung Volume Reduction

INTERVENTIONS:
Biological: Biologic Lung Volume Reduction — 20 mL Hydrogel

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the 20 mL BLVR System in patients with homogeneous emphysema. Patients with upper lobe predominant emphysema initially screened for earlier Phase 2 studies but not enrolled before study enrollment closed are also eligible for participation.

DETAILED DESCRIPTION:
Patients with emphysema currently have limited treatment choices. Many patients are treated with steroids and inhaled medications, which often provide little or no benefit. In recent years, lung volume reduction surgery has become an accepted therapy for advanced emphysema. Lung volume reduction surgery (LVRS) involves the removal of diseased portions of the lung in order to enable the remaining, healthier portions of the lung to function better. LVRS, although effective for many patients, is complicated and is accompanied by substantial morbidity and mortality risk.

Aeris Therapeutics has developed the Biologic Lung Volume Reduction (BLVR) System which is intended to achieve lung volume reduction without surgery and its attendant risks. Patients are treated using a bronchoscope to direct treatment to the most damaged areas of the lung or in the case of homogeneous disease, areas that are less active as shown by the extent of regional blood flow. The treatment delivers a precisely proportioned proprietary mixture of drugs and biologics which, when combined at the treatment site, form a biodegradable hydrogel. The hydrogel acts to reduce lung volume by permanently collapsing and sealing the treated areas of the lung. This provides room within the chest to allow the remaining portions of the lung to function better.

Aeris' BLVR development program has been granted Fast Track designation by the U.S. FDA, and is the subject of ongoing clinical trials designed to investigate the safety and efficacy of the BLVR System as a treatment for patients with advanced heterogeneous (upper lobe predominant) emphysema. Fast Track designation is reserved for drug and biologic development programs that are intended to treat serious or life-threatening conditions and that demonstrate the potential to address unmet medical needs.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of advanced homogeneous or upper lobe predominant emphysema demonstrated by CT scan
* age >/= 40 years
* clinically significant dyspnea
* failure of standard medical therapy (typically inhaled beta agonist & inhaled anticholinergic) to relieve symptoms
* pulmonary function tests within protocol-specified ranges (post bronchodilator FEV1 < 45% predicted & experiencing < 30% or 300 mL improvement using bronchodilator; total lung capacity > 110% predicted; residual volume > 150% predicted)
* 6 Minute Walk Distance >/= 150 m

Exclusion Criteria:

* tobacco use within 4 months of initial visit or during study
* body mass index < 15 kg/m2 or> 35 kg/m2
* clinically significant asthma, chronic bronchitis or bronchiectasis
* allergy or sensitivity to procedural components
* pregnant, lactating or unwilling to use birth control if required
* prior lung volume reduction surgery, lobectomy, pneumonectomy, lung transplant, endotracheal valve placement, airway stent placement or pleurodesis
* comorbid condition that could adversely influence outcomes
* inability to tolerate bronchoscopy under conscious sedation (or anesthesia)
* history of renal infarction or renal failure lung perfusion scan indicating > 20% of blood flow to either upper lung field or 30% total to both upper lung fields if homogeneous emphysema

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
reduction in gas trapping | 12 weeks post treatment

SECONDARY OUTCOMES:
improvement in exercise capacity | 12 weeks post treatment
improvement in expiratory flow | 12 weeks post treatment
improvement in vital capacity | 12 weeks post treatment
improvement in dyspnea sysmptoms | 12 weeks post treatment
improvemnet in respiratory quality of life | 12 weeks post treatment
serious adverse events | through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gotfried, MD, Principal Investigator — Pulmonary Associates, Phoenix, AZ; Mark Dransfield, MD, Principal Investigator — University of Alabama, Birmingham, AL; Gerard Criner, MD, Principal Investigator — Temple University Lung Center, Philadelphia, PA; William Leeds, DO, Principal Investigator — Veritas Clinical Specialties, Topeka, KS; Mark Krasna, MD, Principal Investigator — St Josephs Medical Center, Towson, MD; Thomas Gildea, MD, Principal Investigator — Cleveland Clinic, Cleveland, OH; Sanjiv Tewari, MD, Principal Investigator — Akron Medical Center, Akron, OH; Geoffrey McLennan, MD, Principal Investigator — University of Iowa Hospitals & Clinics, Iowa City, IA
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Veritas Clinical Specialties, Topeka, Kansas
  - St Josephs Medical Center, Towson, Maryland
  - Akron Medical Center, Akron, Ohio
  - Cleveland Clinic Foundation, Pulmonary Allergy & Critical Care Medicine, Cleveland, Ohio
  - Temple University Lung Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Background] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216